CLINICAL TRIAL: NCT00805324
Title: Evaluation of the Efficacy and Safety of Desloratadine Syrup in Children Suffering From Seasonal Allergic Rhinitis With or Without Intermittent Asthma
Brief Title: Study of the Effectiveness and Safety of Desloratadine (Aerius) Syrup in Children With Hayfever With or Without Asthma (P03472)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03472
Record Dates: First submitted 2008-12-05; First posted 2008-12-09 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal; Asthma
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Asthma | interventions — desloratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Desloratadine

INTERVENTIONS:
Drug: Desloratadine — desloratadine syrup; 5.0 mL once daily for 28 days
  Other Names: Clarinex; Aerius; SCH 34117; descarboethoxyloratadine

SUMMARY:
The purpose of this study was to test the effectiveness and safety of desloratadine (Aerius) syrup in children with hayfever with or without asthma. Patients took desloratadine syrup once a day for 28 days. Once a week, the doctor measured the patient's hayfever symptoms. The doctor also rated how much relief the patient got from treatment and recorded any side effects.

ELIGIBILITY:
Inclusion Criteria:

* Children must be >= 6 to < 12 years of age of either sex and any race.
* Children's parent(s) or legal representative(s) must demonstrate their willingness to participate in the study and comply with its procedures by signing an informed consent
* Children must be free of any clinically significant disease (other than SAR) that would interfere with study evaluations
* Children's parent(s) or legal representative(s) must understand and be able to adhere to dosing and visit schedules, agree to report concomitant medications and adverse events to the Investigator or designee
* The diagnosis of seasonal allergic rhinitis with or without intermittent asthma will be assessed by:

  * Clinical history of sneezing, rhinorrhea (nasal discharge/running nose or post-nasal drip), nasal stuffiness/congestion and nasal itching and non-nasal symptoms (eye symptoms) as itching, burning, tearing and redness, during the previous pollen season
  * Ascertained skin prick positivity (or RAST positivity) to one of the following: grasses, parietaria, birch, hazelnut (the skin test has to be performed within the last year)
* Children must be clinically symptomatic with SAR at Visit 1 (day 1): the total (nasal + non nasal) symptoms score must be >= 8 with a nasal congestion score of >= 2, and the non-nasal symptoms severity score must be >= 2
* Asthma symptoms (wheezing, cough, difficulty breathing, chest tightness) will be evaluated at visit 1 (day 1) and graded only for child with concomitant asthma

Exclusion Criteria:

* Children who have not observed the designated washout periods for any of the prohibited medications

  * Children with persistent asthma (mild, moderate or severe) or perennial allergic rhinitis (PAR)
* Children with rhinitis medicamentosa
* Children who have had an upper respiratory tract or sinus infection that required antibiotic therapy within 14 days prior to Visit 1 (day 1), or children who have had a viral upper respiratory infection within 7 days prior to Visit 1 (day 1)
* Children who have nasal structural abnormalities, including nasal polyps and marked septal deviation, that significantly interfere with nasal airflow
* Children who, in the opinion of the Investigator, are dependent upon nasal, oral or ocular decongestants, nasal topical antihistamines, or nasal steroids
* Children with a history of hypersensitivity to desloratadine or any of its excipients
* Children who have any current clinically significant metabolic, cardiovascular, hepatic, renal, immunologic, neurologic, hematologic, gastrointestinal, cerebrovascular or respiratory disease, or any other disorder which, in the judgment of the Investigator, may interfere with the study evaluations or affect subject safety
* A known lack of response to H1-antihistamines

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2003-05; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Demonstration of the efficacy of desloratadine in relieving the total nasal/non-nasal symptoms of seasonal allergic rhinitis | Baseline, Day 8, Day 15, Day 29

SECONDARY OUTCOMES:
To demonstrate that the Global Therapeutic Response is correlated with the degree of improvement of the total nasal/non-nasal symptoms severity score | Day 8, Day 15, Day 29
To evaluate the number of adverse events during the therapy | Day 8, Day 15, and Day 29

REFERENCES:
- [Result] Rossi GA, Tosca MA, Passalacqua G, Bianchi B, Le Grazie C, Canonica GW. Evidence of desloratadine syrup efficacy and tolerability in children with pollen-induced allergic rhinitis. Allergy. 2005 Mar;60(3):416-7. doi: 10.1111/j.1398-9995.2005.00714.x. No abstract available. PMID 15679739